CLINICAL TRIAL: NCT00244517
Title: The Effects of Remifentanil, Sevoflurane, Isoflurane and Desflurane on Left Ventricular Diastolic Function in Humans
Brief Title: DIAFAX I+II-Effects of Inhalative Anesthetics on Left Ventricular Diastolic Function
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Part II was not performed as we could not include enough patients fulfilling the inclusion criteria.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Prof. Dr. M. Seeberger, Head of Cardiothoracic Anesthesia, University Hospital Basel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 225/03
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Young Healthy Adults; Ventricular Dysfunction
Keywords: ventricular function; diastolic function; inhalative anaesthetics
MeSH Terms: conditions — Ventricular Dysfunction | interventions — Sevoflurane; Isoflurane; Desflurane; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Active Comparator): Isoflurane (only in part I)
  Interventions: Drug: TTE measurements under anesthesia with sevoflurane, isoflurane, desflurane, and remifentanyl; Drug: Sevoflurane, Isoflurane, Desflurane
- II (Active Comparator): Sevoflurane
  Interventions: Drug: TTE measurements under anesthesia with sevoflurane, isoflurane, desflurane, and remifentanyl; Drug: Sevoflurane, Isoflurane, Desflurane
- III (Active Comparator): Desflurane
  Interventions: Drug: TTE measurements under anesthesia with sevoflurane, isoflurane, desflurane, and remifentanyl; Drug: Sevoflurane, Isoflurane, Desflurane

INTERVENTIONS:
Drug: TTE measurements under anesthesia with sevoflurane, isoflurane, desflurane, and remifentanyl — TTE measurements were performed during remifentanil 2 ng/ml TCI end-organ concentration, 1 MAC of either anesthetic gas under spontaneous ventilation and 1 MAC of either anesthetic under IPPV
Drug: Sevoflurane, Isoflurane, Desflurane — 1 MAC

SUMMARY:
Anaesthetics may impair the diastolic function of the heart, but the importance of this finding for patients has not been sufficiently examined. Specially the effects on diastolic function in patients with diastolic dysfunction has to be determined. The aim of this study is to examine the effect of isoflurane (only part I), sevoflurane and desflurane (part I+II) on the diastolic left ventricular function by doppler echocardiography.

DETAILED DESCRIPTION:
In part I, 60 healthy young subjects free from cardiovascular disease will be examined. In part II, 50 patients with impaired diastolic but preserved systolic function, i.e., patients with arterial hypertension and ejection fraction > 50%. Doppler echocardiography will be performed at baseline before induction of anaesthesia, during anaesthesia in the spontaneously breathing patient, and in the mechanically ventilated patient.

ELIGIBILITY:
Inclusion Criteria:

* part I: 18- to 50-year-old patients undergoing surgical procedures under general anesthesia
* part II: 50-years-old patients or older with arterial hypertension under chronic antihypertensive medication subsequently undergoing surgical procedures under general anesthesia, EF >50%

Exclusion Criteria:

* part I: any cardiac or pulmonary disease, any medication with cardiovascular effects or side effects, body mass index > 30 kg/m2, esophageal reflux, emergency
* part II: History of myocardial infarction or coronary revascularization, severe lung disease, body mass index > 30 kg/m2, esophageal reflux, emergency

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To determine the effect of the opiate remifentanil and of the inhalative anaesthetics isoflurane (only part I), sevoflurane and desflurane on the diastolic function of the left ventricle in healthy young adults, and in patients with diastolic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Seeberger, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, CH, Switzerland